CLINICAL TRIAL: NCT01592344
Title: Prospective, Multi-Center, Randomized, Double-Blinded, Study to Assess Safety and Efficacy of the Bioness® StimRouter™ Neuromodulation System in Patients With Chronic Pain of Peripheral Nerve Origin
Brief Title: Bioness® StimRouter™ Neuromodulation System for Chronic Pain Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioness Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CP-STMR11-001
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Pain
Keywords: Chronic pain; peripheral nerve; neuralgia; somatosensory nervous system
MeSH Terms: conditions — Chronic Pain; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- StimRouter - active stimulation (Experimental): StimRouter- active electrical stimulation is applied transdermally to a targeted peripheral nerve. This is accomplished via a fully implanted StimRouter lead that receives energy from a rechargeable programmed external pulse transmitter (EPT) with attached gel electrodes. The EPT receives radio frequency (RF) commands from a Patient Programmer. A StimRouter Clinician Programmer is used to program the StimRouter EPT and Patient Programmer. Up to eight stimulation programs may be saved on a Patient Programmer for on-demand selection by the study patient.
  Interventions: Device: StimRouter - active stimulation
- StimRouter - Control (Sham Comparator): StimRouter- Electrical stimulation is withheld from the targeted peripheral nerve after fully implanting the StimRouter lead. The rechargeable programmed external pulse transmitter (EPT) with attached gel electrodes is placed for transdermal stimulation but no stimulation is delivered. The EPT which normally receives radio frequency (RF) commands from a Patient Programmer is not activated. A StimRouter Clinician Programmer is used to program the StimRouter EPT and Patient Programmer such that no stimulation occurs in the Control Arm of the study.
  Interventions: Device: StimRouter - Control

INTERVENTIONS:
Device: StimRouter - active stimulation — The stimulation program settings for this arm are as follows:
  Stim Settings
  * Waveform: Symmetric or Asymmetric
  * Phase Duration: 100-250 µsec
  * Pulse Rate: 50-100 Hz
  * Intensity: 0-30mA Time Settings
  * Constant Stim: On
  * Total Time: 6 hour
  Other Names: Bioness® StimRouter™ Neuromodulation System
  Arms: StimRouter - active stimulation
Device: StimRouter - Control — The stimulation program settings for this arm are as follows:
  Stim Settings
  * Waveform: Symmetric or Asymmetric
  * Phase Duration: 200 µsec
  * Pulse Rate: 1 Hz
  * Intensity: 0 mA Time Settings
  * Constant Stim: On
  * Total Time: 6 hour
  Other Names: Bioness® StimRouter™ Neuromodulation System
  Arms: StimRouter - Control

SUMMARY:
The purpose of this study is to investigate whether the StimRouter (SR) electrical stimulation therapy leads to clinically important pain relief in patients with chronic intractable pain of peripheral nerve origin after three months of treatment. At the same time, this study will gather information on side effects associated with the StimRouter electrical stimulation therapy.

DETAILED DESCRIPTION:
Ninety (minimum) up to one hundred twenty-six (126) adult (≥ 22 years) subjects who have severe intractable chronic pain of peripheral nerve origin associated with post traumatic/post surgical neuralgia persisting for 3 months or longer and an average chronic pain level of at least 5 on a 0-10 numeric rating scale, where such pain is attributable to a lesion or disease of the somatosensory nervous system, will be recruited from U.S. outpatient physical medicine and rehabilitation clinics.

After screening, subjects who were confirmed to be eligible for the study and provided informed consent will have a pain level assessment period for approximately one week then come back for the Baseline/Implantation visit. Subjects will be trained on and required to complete a patient diary of pain intensity level for at least 7 consecutive days prior to baseline. The randomization and programming will take place approximately two weeks after implantation. Subjects in the treatment group will receive electrical stimulation and pain medication. In contrast, subjects in the parallel control group will receive control stimulation and pain medication.

The plan is to have the parallel portion of the study run for approximately 12 weeks (or 3 months) after randomization for efficacy analysis. Subjects in the control group will be allowed to cross over to the treatment group for nine months of electrical stimulation; the subjects in the treatment group will have nine additional months of stimulation treatment such that safety data will be collected throughout a full twelve month period on all available subjects. While the end of the study is approximately 12 months after randomization, as previously stated, the efficacy analyses will be based on the data collected at the end of the 3-month follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 22 years) suitable for an implanted electrode for pain relief.
2. Subjects who are able to give informed consent and to understand and comply with study requirements.
3. Subjects who have severe intractable chronic pain of peripheral nerve origin associated with post traumatic/post surgical neuralgia for ≥ 3 months (i.e., intractable to pain medication).
4. Subjects who are able to tolerate skin surface stimulation (TENS).
5. Subjects who have a worst chronic pain level in the last 24 hours ≥ 5/10 (on 0-10 NRS) where such pain is attributable to a lesion or disease of the somatosensory nervous system.
6. Subjects who are on a stable dose of pain medications for at least four weeks prior to screening and willing and able to maintain an equivalent dosage of their current pain medications from randomization to 3-month follow-up.

Exclusion Criteria:

1. Subjects who are not willing and able to maintain stable dosages of their pain medications from randomization to 3-month follow-up.
2. Subjects with a pain condition that could be confused with their peripheral neuropathic pain or that is more severe than their peripheral neuropathic pain.
3. Subjects who, for implantation in the trunk, have an implanted demand-type cardiac pacemaker or defibrillator.
4. Subjects who have a metal implant in the area for StimRouter implantation without Sponsor approval. Maintain a minimum separation distance of 6 inches (15 cm) between the StimRouter system and all other active implanted devices and metallic implants.
5. Subjects who require, or are likely to require, diathermy at the implant site.
6. Subjects who require, or are likely to require, therapeutic ultrasound at the implant site.
7. Subjects who have a cancerous lesion present near the target stimulation point or near to where the StimRouter user patch will adhere.
8. Subjects who are known or suspected to have a nickel allergy.
9. Subjects with bleeding disorders or active anticoagulation that cannot be stopped for a few days close to the time of the surgical procedure.
10. Subjects who decline to provide written consent or follow-up.
11. Subjects who are pregnant, plan on becoming pregnant, or are breastfeeding during the study period. Subjects who are female of child-bearing potential must have a negative pregnancy test at baseline visit and, if sexually active, must be using a medically acceptable method of contraception for the duration of the study participation.
12. Subjects who have an active systemic infection or are immunocompromised.
13. Subjects who have an active or existing skin disorder or irritation, which, at the physician's discretion, precludes the use of skin gel electrodes.
14. Subjects who currently require or are likely to require Magnetic Resonance Imaging (MRI) within the MRI exclusion zone: the entire StimRouter lead must be at least 50 cm from the center of the MR system's bore (the iso-center) and at least 16 cm outside of the MR coil measured from the edge of the MR coil.
15. Subjects who have a history of adverse reactions to local anesthetic (e.g., lidocaine).
16. Subjects who are participating in any other study that could affect the outcome of the StimRouter study, such as a spinal stimulation study, without Sponsor approval.
17. Subjects who are in litigation or who have pending or an active worker's compensation claim.
18. Subjects with less than one year of life expectancy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linh Nguyen, MS, Study Director — Bioness Inc; Ramsin Benyamin, M.D., Principal Investigator — Millennium Pain Center; Timothy Deer, M.D., Study Chair — Center for Pain Relief, St. Francis Hospital
Locations (13):
- United States (13):
  - Arizona Pain Specialists, Scottsdale, Arizona
  - Neurovations, Napa, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - The Spine Institute, Center for Spinal Restoration, Santa Monica, California
  - Holy Cross Orthopedic Institute, Fort Lauderdale, Florida
  - Shands Jacksonville Medical Center, Dept of Neurology Research, Jacksonville, Florida
  - Millennium Pain Center, Bloomington, Illinois
  - Premier Pain Centers, LLC, Shrewsbury, New Jersey
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Virginia Mason Medical Center, Seattle, Washington
  - Center for Pain Relief, St. Francis Hospital, Charleston, West Virginia
  - The Center for Pain Relief at St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- See also: MedlinePlus related topics: Chronic pain — http://www.nlm.nih.gov/medlineplus/chronicpain.html
- See also: US FDA Recourses — http://clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Stimulation Treatment: Subjects implanted with the StimRouter lead and randomized to receive active stimulation.
- Control: Subjects implanted with the StimRouter lead and randomized to receive no electrical stimulation.
Period: Overall Study
Arm/Group | Active Stimulation Treatment | Control
Started | 45 | 49
Completed | 41 | 44
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — not available at primary outcome visit | 2 | 4

BASELINE CHARACTERISTICS:
Population: Adults having severe intractable chronic pain of peripheral nerve origin were enrolled and all were included in the 94 intent-to-treat analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation Treatment | Control | Total
Number analyzed (Participants) | 45 | 49 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (10.0) | 53.2 (12.1) | 53.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 45 | 49 | 94

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI): Number of Participants With a Pain Reduction of Greater Than or Equal to 30%
Description: The average pain at rest was assessed using a numerical (0-10) rating scale (NRS) on the Brief Pain Inventory (BPI) Short Form (SF). A higher score indicates worse pain (10=worst pain imaginable) and zero indicates 'no pain at all'. A pain reduction of greater than or equal to 30% on the NRS was considered to be clinically relevant.
Time Frame: Baseline and at 3-month follow-up.
Population: Intent to treat (ITT) population was analyzed.
Measure: Number; unit: participants
Groups:
- StimRouter - Active Stimulation: StimRouter- active electrical stimulation is applied transdermally to a targeted peripheral nerve. This is accomplished via a fully implanted StimRouter lead that receives energy from a rechargeable programmed external pulse transmitter (EPT) with attached gel electrodes. The EPT receives radio frequency (RF) commands from a Patient Programmer. A StimRouter Clinician Programmer is used to program the StimRouter EPT and Patient Programmer. Up to eight stimulation programs may be saved on a Patient Programmer for on-demand selection by the study patient.
  StimRouter - active stimulation: The stimulation program settings for this arm are as follows:
  Stim Settings
  * Waveform: Symmetric or Asymmetric
  * Phase Duration: 100-250 µsec
  * Pulse Rate: 50-100 Hz
  * Intensity: 0-30mA Time Settings
  * Constant Stim: On
  * Total Time: 6 hour
- StimRouter - Control: StimRouter- Electrical stimulation is withheld from the targeted peripheral nerve after fully implanting the StimRouter lead. The rechargeable programmed external pulse transmitter (EPT) with attached gel electrodes is placed for transdermal stimulation but no stimulation is delivered. The EPT which normally receives radio frequency (RF) commands from a Patient Programmer is not activated. A StimRouter Clinician Programmer is used to program the StimRouter EPT and Patient Programmer such that no stimulation occurs in the Control Arm of the study.
  StimRouter - Control: The stimulation program settings for this arm are as follows:
  Stim Settings
  * Waveform: Symmetric or Asymmetric
  * Phase Duration: 200 µsec
  * Pulse Rate: 1 Hz
  * Intensity: 0 mA Time Settings
  * Constant Stim: On
  * Total Time: 6 hour
Arm/Group | StimRouter - Active Stimulation | StimRouter - Control
Number analyzed (Participants) | 45 | 49
participants | 17 | 5
Statistical Analysis 1: Comparison: StimRouter - Active Stimulation vs StimRouter - Control; Test type: Superiority or Other; p = 0.0048, Cochran-Mantel-Haenszel

2. Secondary Outcome: Patient Global Impression of Improvement With Treatment Will be Assessed Using the Patient Global Impression of Change Scale (PGIC).
Description: Patient Global Impression of Change in activity limitations, symptoms, emotions and overall life quality related to their painful condition (Range 1 to 7, with 1 indicating no change and 7 indicating a great deal better/considerable improvement).
Time Frame: at 3 month follow-up
Population: All patients who completed the 3 month Global Impression of Change questionnaire were included. Four patients in each study arm failed to complete the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StimRouter - Active Stimulation | StimRouter - Control
Number analyzed (Participants) | 41 | 45
units on a scale | 4.8 (1.5) | 2.5 (1.9)
Statistical Analysis 1: Comparison: StimRouter - Active Stimulation vs StimRouter - Control; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Worst Pain in the Last 24 Hours Will be Assessed Using 7-day Patient Pain Diary Scores for BPI SF #3.
Description: Worst pain in the last 24 hours assessed using 7-day patient pain diary scores for BPI ranging from 0 to 10, with 0 indicating no pain and 10 indicating "pain as bad as you can imagine". Change from baseline to Month 3 was compared.
Time Frame: at baseline and 3 month follow-up
Population: All available data were analyzed from both treatment arms.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StimRouter - Active Stimulation | StimRouter - Control
Number analyzed (Participants) | 41 | 45
units on a scale | -2.4 (2.3) | -0.3 (1.6)
Statistical Analysis 1: Comparison: StimRouter - Active Stimulation vs StimRouter - Control; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Patient Satisfaction Will be Assessed Using a Patient Satisfaction Survey
Description: Patient satisfaction with the StimRouter System was rated on a numerical rating scale (range 0 to 10), with 0 indicating not satisfied at all and 10 indicating completely satisfied.
Time Frame: at the 3-month follow-up
Population: All subjects who completed the survey at Month 3 were included in this analysis. Four subjects in each study arm (4/45 Treatment; 4/49 Control) failed to complete the satisfaction survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | StimRouter - Active Stimulation | StimRouter - Control
Number analyzed (Participants) | 41 | 45
units on a scale | 7.3 (2.9) | 3.0 (3.6)
Statistical Analysis 1: Comparison: StimRouter - Active Stimulation vs StimRouter - Control; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were reported throughout the one year study period.
Description: No device related serious adverse events were reported.
Groups:
- StimRouter Active Stimulation: The stimulation program settings for the active stimulation arm are as follows:
  Stim Settings
  * Waveform: Symmetric or Asymmetric
  * Phase Duration: 100-250 µsec
  * Pulse Rate: 50-100 Hz
  * Intensity: 0-30mA Time Settings
  * Constant Stim: On
  * Total Time: 6 hour
- StimRouter Control: The stimulation program settings for the control arm are as follows:
  Stim Settings
  * Waveform: Symmetric or Asymmetric
  * Phase Duration: 200 µsec
  * Pulse Rate: 1 Hz
  * Intensity: 0 mA Time Settings
  * Constant Stim: On
  * Total Time: 6 hour
Arm/Group | StimRouter Active Stimulation | StimRouter Control
Serious Adverse Events (participants affected / at risk) | 9/45 | 11/49
Other Adverse Events (participants affected / at risk) | 19/45 | 16/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StimRouter Active Stimulation (N=45) | StimRouter Control (N=49)
heart arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) — Unrelated to device
Kidney failure and bladder tumor (Renal and urinary disorders) | 3 (4) | 0 (0) — unrelated to device
gall bladder (Hepatobiliary disorders) | 1 (1) | 2 (2) — cholelithiasis and cholecystectomy not device related
Bone fracture, instability, compromise (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (3) — Knee replacement, rotator cuff repair, spine instability/leak, bone fracture all unrelated to device
Respiratory issues (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — unrelated to device: pneumonia, breathing problems
Digestive issues (Gastrointestinal disorders) | 0 (0) | 2 (2) — diverticulitis not device related
dermatological issues (Infections and infestations) | 1 (1) | 2 (2) — unrelated abscess, cellulitis, infection,
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — unrelated dehydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StimRouter Active Stimulation (N=45) | StimRouter Control (N=49)
Localized pain irritation to patch/wound site (Skin and subcutaneous tissue disorders) | 15 (33) | 16 (26)
Gastrointestinal (Gastrointestinal disorders) | 3 (5) | 3 (5) — diarrhea, diverticulitis, nausea
renal (Renal and urinary disorders) | 3 (3) | 2 (2) — kidney stone, urinary tract infection, kidney function
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) — flu, cough
Infection (Infections and infestations) | 1 (1) | 2 (3) — sinusitis
Psychiatric (Psychiatric disorders) | 0 | 1 (2) — confusion, dementia
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (6) | 7 (18) — Joint spine issues
Fall/bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) — Falling due to frailty
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Delayed ejaculation
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
headache (General disorders) | 2 (4) | 0 (0)
Medicine wthdrawn in error (General disorders) | 1 (1) | 0 (0)
Lead exposure (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) — lead implanted too superficially, skin scratched by patient until lead became exposed requiring repositioning of lead

LIMITATIONS AND CAVEATS:
The device was designed for treatment of mononeuritis excluding the face. For this reason, mononeuropathies of the face were excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less